CLINICAL TRIAL: NCT07076303
Title: A Prospective Study on the Efficacy of Direct Selective Laser Trabeculoplasty (DSLT) in Achieving >20% Intraocular Pressure (IOP) Reduction Without Medications at 6 Months in Naive, Untreated Glaucoma Patients
Status: Recruiting | Type: Observational
Sponsor: Brian Shafer (Other)
Responsible Party: Sponsor-Investigator, Brian Shafer, Ophthalmologist, Shafer Vision Institute
Organization: Shafer Vision Institute (Other)
Other Study IDs: 95532219
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Primary Open Angle Glaucoma; Glaucoma; Primary Open Angle Glaucoma or Ocular Hypertension
Keywords: glaucoma; primary open angle glaucoma; direct SLT; SLT; selective laser trabeculoplasty
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Primary Open Angle Glaucoma or Ocular Hypertension: Subjects with primary open angle glaucoma or ocular hypertension with baseline IOPs greater than 21mmHg.
  Interventions: Device: Direct Selective Laser Trabuloplasty

INTERVENTIONS:
Device: Direct Selective Laser Trabuloplasty — Eligible participants will undergo the DSLT procedure to facilitate controlled aqueous outflow. DSLT will consist of 120 shots, 400 µm spot size, energy 1.4-1.8 mJ delivered at the limbus over 2.4 seconds
  Other Names: DSLT; Eagle DSLT

SUMMARY:
Background

Glaucoma is a progressive optic neuropathy characterized by elevated intraocular pressure (IOP), leading to irreversible vision loss. Current treatment strategies often involve medications, which can be challenging for patients due to adherence issues and side effects. Direct Selective Laser Trabeculoplasty (DSLT) represents a potential surgical alternative for managing IOP in patients with naive, untreated glaucoma. This study aims to evaluate the efficacy of DSLT in achieving significant IOP reduction without the need for postoperative medications.

Unmet Medical Need:

Overview of DSLT

Direct Selective Laser Trabeculoplasty (DSLT) is an emerging technology in glaucoma management that combines laser techniques to reduce intraocular pressure (IOP). While it works off the auspices of a previous technology (SLT), the method of delivery is significantly different.

Current Research Landscape

Most existing studies focus on patients who have already received other forms of treatment or who have more advanced glaucoma. This creates an unmet need to evaluate how DSLT can be effectively integrated into the management of patients at the very beginning of their glaucoma journey. Understanding its efficacy in this population is crucial for establishing best practices and improving long-term outcomes.

Interventional Glaucoma Management vs. Standard of Care

Standard of care for newly diagnosed glaucoma typically involves medications, such as topical prostaglandin analogs, which can have side effects and may not be effective for all patients. In contrast, interventional glaucoma management-such as DSLT-offers a potentially more direct approach to lowering IOP without the need for ongoing medication. Investigating DSLT in this context could lead to a paradigm shift in how newly diagnosed patients are managed, reducing their reliance on medications and potentially improving adherence and quality of life.

Conclusion

Addressing this research gap will not only help clarify the role of DSLT in early glaucoma management but could also enhance patient outcomes and guide future treatment protocols. Focusing on newly diagnosed patients is essential for determining the long-term benefits and risks associated with this innovative technology.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older:

Participants must be adults, aged 18 years or older, to ensure they are capable of providing informed consent and to focus on adult-onset glaucoma. This age threshold allows the study to target a population where open-angle glaucoma typically manifests, avoiding potential variations in outcomes that might arise in younger populations with different types of ocular conditions.

Diagnosis of naive, untreated open-angle glaucoma or similar conditions:

The study is restricted to individuals who have been newly diagnosed with primary open-angle glaucoma and have not yet received any form of treatment, either pharmacological or surgical. This ensures that the effects of DSLT (Direct Selective Laser Trabeculoplasty) are evaluated without the confounding influence of prior treatments.

Other similar conditions may include ocular hypertension or other early-stage glaucomatous conditions where IOP reduction is indicated (ie: pigment dispersion syndrome/glaucoma and pseudoexfoliation). This broadens the inclusion slightly to capture patients with conditions that have a similar disease mechanism and treatment goal, without including those with more complex or mixed forms of glaucoma.

Exclusion Criteria:

Previous glaucoma surgeries/interventions:

Patients who have undergone prior glaucoma-related surgeries (e.g., trabeculectomy, laser trabeculoplasty, or shunt procedures) or received other significant glaucoma interventions (such as long-term glaucoma medication use) are excluded. This criterion ensures the study evaluates the effect of DSLT in a treatment-naive population. Prior surgeries or interventions could bias the results by introducing variability in eye physiology, making it difficult to attribute outcomes solely to DSLT.

Secondary glaucoma or other significant ocular conditions:

Patients with secondary forms of glaucoma, such as angle-closure glaucoma, neovascular glaucoma, or glaucoma resulting from trauma or other systemic diseases, are excluded. These conditions often have different pathophysiological mechanisms, which could lead to varied responses to DSLT.

Other significant ocular conditions that could interfere with the study include advanced cataracts, retinal diseases (e.g., age-related macular degeneration), or any condition that might complicate the assessment of intraocular pressure (IOP) or visual function. Excluding these conditions ensures a clearer evaluation of DSLT's effects on open-angle glaucoma without interference from unrelated ocular abnormalities.

3. Patients who are unable to fixate their head and/or eyes, such as patients suffering from uncontrolled nystagmus, tremors, or similar conditions.

4. Patients with a pupil that cannot constrict to a diameter of 4 mm or less.

In summary, these criteria focus on a specific and controlled population of treatment-naive glaucoma patients to provide a clean evaluation of the effectiveness and safety of DSLT, while excluding individuals whose prior treatments or other conditions could skew the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older who have primary open angle glaucoma or ocular hypertension who are treatment naïve.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2002-03-11 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent Reduction in IOP from baseline at 6 months | 6 months
  Percent Reduction in IOP from baseline at 6 months

SECONDARY OUTCOMES:
Percentage of Eyes Achieving ≥ 20% Reduction in IOP at 6 months | 6 months
  The success rate of IOP reduction at 6 months, where success is defined as % of eyes achieving ≥20% reduction from baseline pre-treatment IOP.
IOP reduction from baseline at 1 and 3 months | 3 months
  Percentage IOP reduction from baseline at 1 and 3 months
Rate of Secondary Interventions at 6 months | 6 months
  The rate of secondary interventions (e.g., additional treatment or procedures) at 6 months post-DSLT.

CONTACTS AND LOCATIONS:
Locations (1):
- Shafer Vision Institute, Plymouth Meeting, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The IPD is kept private at Shafer Vision Institute and is not available for outside access.

REFERENCES:
- [Background] Congdon N, Azuara-Blanco A, Solberg Y, Traverso CE, Iester M, Cutolo CA, Bagnis A, Aung T, Fudemberg SJ, Lindstrom R, Samuelson T, Singh K, Blumenthal EZ, Gazzard G; GLAUrious study group. Direct selective laser trabeculoplasty in open angle glaucoma study design: a multicentre, randomised, controlled, investigator-masked trial (GLAUrious). Br J Ophthalmol. 2023 Jan;107(1):62-65. doi: 10.1136/bjophthalmol-2021-319379. Epub 2021 Aug 25. PMID 34433548
- [Background] Goldenfeld M, Belkin M, Dobkin-Bekman M, Sacks Z, Blum Meirovitch S, Geffen N, Leshno A, Skaat A. Automated Direct Selective Laser Trabeculoplasty: First Prospective Clinical Trial. Transl Vis Sci Technol. 2021 Mar 1;10(3):5. doi: 10.1167/tvst.10.3.5. PMID 34003939